CLINICAL TRIAL: NCT03988569
Title: Enhanced Consent and Preparedness for Surgery (ECAPS) Trial
Brief Title: Enhanced Consent and Preparedness for Surgery Trial
Acronym: ECAPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Responsible Party: Principal Investigator, Marian G. Acevedo Alvarez, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 212237
Record Dates: First submitted 2019-06-03; First posted 2019-06-17 (Actual); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Stress Urinary Incontinence; Urge Incontinence; Pelvic Organ Prolapse
MeSH Terms: conditions — Urinary Incontinence, Stress; Urinary Incontinence, Urge; Pelvic Organ Prolapse

STUDY DESIGN:
Intervention Model Description: the proposed study is to test the null hypothesis that there is no difference in surgical preparedness between women who receive a standard surgical consent for pelvic reconstructive surgery (control) and those who receive a standard surgical consent that is enhanced with an audiovisual decision aid (treatment) for the same surgery. Equivalently, the null hypothesis is that the odds ratio is 1.00.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): Will view audiovisual decision aid (AVDA) and then have opportunity for questions with physician before signing consent forms
  Interventions: Other: audiovisual decision aid
- Control Group (No Intervention): Will undergo standard verbal informed consent with physician before signing consent forms

INTERVENTIONS:
Other: audiovisual decision aid — Will view AVDA and then have opportunity for questions with physician before signing consent forms
  Arms: Intervention Group

SUMMARY:
To develop an audiovisual decision aid (AVDA) to improve the informed consent process. The investigators aim to examine the impact of a comprehensible AVDA that is written below the 8th grade reading level. The AVDA would be used for surgical consent compared to traditional verbal consent. Additionally, the investigators plan to determine whether this effect varies across the measured levels of health literacy of our patients.

DETAILED DESCRIPTION:
To address the limitations of consent, interventions have been developed to improve the quality of information provided to patients including written pamphlets, videos, and websites. Such interventions have been called decision aids. Decision aids may promote informed consent through greater knowledge and consistency of personal values or attitudes with an enacted choice. Providing adequate information increases satisfaction, more rapid symptom resolution, reduced emotional distress, reduced use of analgesia, and possibly shorter hospital admissions. Cochrane reviews have established that audiovisual decision aids enhance informed surgical consent, yet little data exists about the benefits of such aids in Female Pelvic Medicine and Reconstructive Surgery (FPMRS)4.

ELIGIBILITY:
Inclusion Criteria:

* Patients electing for surgical intervention of pelvic organ prolapse, stress urinary incontinence, urgency urinary incontinence by treating physicians in the Female Pelvic Medicine & Reconstructive Surgery.

Exclusion Criteria:

* Patients ≤ 18 years old
* Non-English speaking patients
* Patients with video or audio impairments who are unable to view the AVDA

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2024-02-22 (Actual)

PRIMARY OUTCOMES:
Preparedness for surgery | Day 0
  To compare the odds of higher agreement between patients assigned to receive enhanced audiovisual aided consent versus standard consent on the question "Overall, I feel prepared for my upcoming surgery". This item is asked on day of consent and patients respond using a six-point Likert scale ranging from 0 (Strongly disagree) to 5 (Strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Marian G Acevedo-Alvarez, MD, Principal Investigator — Loyola Medical Center
Locations (1):
- Loyola Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vos IML, Schermer MHN, Bolt ILLE. Recent insights into decision-making and their implications for informed consent. J Med Ethics. 2018 Nov;44(11):734-738. doi: 10.1136/medethics-2018-104884. Epub 2018 Jul 21. PMID 30032106
- [Background] Weiss BD, Blanchard JS, McGee DL, Hart G, Warren B, Burgoon M, Smith KJ. Illiteracy among Medicaid recipients and its relationship to health care costs. J Health Care Poor Underserved. 1994;5(2):99-111. doi: 10.1353/hpu.2010.0272. PMID 8043732
- [Background] Institute of Medicine (US) Committee on Health Literacy; Nielsen-Bohlman L, Panzer AM, Kindig DA, editors. Health Literacy: A Prescription to End Confusion. Washington (DC): National Academies Press (US); 2004. Available from http://www.ncbi.nlm.nih.gov/books/NBK216032/ PMID 25009856
- [Background] Baker DW, Williams MV, Parker RM, Gazmararian JA, Nurss J. Development of a brief test to measure functional health literacy. Patient Educ Couns. 1999 Sep;38(1):33-42. doi: 10.1016/s0738-3991(98)00116-5. PMID 14528569